CLINICAL TRIAL: NCT05150080
Title: Early Identification and Evaluation of the Cardiotoxicity of Cyclophosphamide in Hematopoietic Stem Cell Transplantation : Based on Spot Tracking Ultrasound
Brief Title: Early Identification and Evaluation of Cyclophosphamide Cardiotoxicity
Acronym: EIECC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kai Mu (Other)
Responsible Party: Sponsor-Investigator, Kai Mu, Clinical Research Assistant, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QianfoshanH-210118
Record Dates: First submitted 2021-11-27; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Cardio-oncology; Hematopoietic Stem Cell Transplantation; Cardiotoxicity; Cyclophosphamide; Echocardiography
Keywords: Cardio-oncology; Speckle tracking echocardiography
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardiotoxicity: subjects with heart failure, coronary artery disease, valvular heart disease, arrhythmia, hypertension, thromboembolic disease, peripheral vascular disease and stroke, pulmonary hypertension and pericardial disease after hematopoietic stem cell transplantation.
- non-cardiotoxicity: subjects with on heart failure, coronary artery disease, valvular heart disease, arrhythmia, hypertension, thromboembolic disease, peripheral vascular disease and stroke, pulmonary hypertension and pericardial disease after hematopoietic stem cell transplantation.

SUMMARY:
Hematopoietic stem cell transplantation is an important method for the treatment of hematological diseases and cyclophosphamide is a commonly used chemotherapeutic agent for transplant pretreatment. The incidence of severe cardiovascular events after high-dose cyclophosphamide exposure ranges from 7% to 28% with mortality from 11% to 43%. Thus, an non-invasive, sensitive and reliable method in detecting cardiac function is significant to balance the cardiac risk and the potential cancer treatment benefits. In previous studies, we demonstrated that strain values analyzed by speckle tracking echocardiography decreased significantly after high-dose cyclophosphamide exposure, even though left ventricular ejection fraction remained stable and within normal range. We follow up the hematopoietic cell transplantation patients with cyclophosphamide: to analyze the cut-off values of the parameters of speckle tracking multilayer analysis in predicting early cardiotoxicity induced by cyclophosphamide; to detect the cut-off values of the plasma miRNAs levels in predicting early cardiotoxicity induced by anthracycline.

The purpose of our study is to find out non-invasive, reliable and sensitive echocardiographic parameters and plasma biomarkers for early detection and prediction cyclophosphamide -induced cardiac toxicity and to be helpful to target patients at high risk of cardiotoxicity, who could benefit from closer monitoring or earlier initiation of cardioprotective therapy.

DETAILED DESCRIPTION:
After obtaining the informed consent of the research subjects, collect the following data of the research subjects: demographic information, clinical symptoms, family history and clinical diagnosis. Patients were tested for troponin, atrial natriuretic peptide, concurrent conventional electrocardiogram, conventional echocardiogram, speckle tracking echocardiography at spots 1 day before cyclophosphamide treatment, 2 days after cyclophosphamide infusion, and 10 days after cyclophosphamide infusion. ethylenediaminetetraacetic acid anticoagulated whole blood were saved and extract the blood cells from the sample bank and freeze them for RNA sequencing. The two-dimensional cardiac ultrasound image acquisition complies with the guidelines of the American Echocardiography Association, and the two-dimensional speckle tracking echocardiography acquisition is 4 cardiac cycles. If a cardiotoxic event occurs during this period, an electrocardiogram, conventional echocardiogram, and speckle tracking echocardiography should be performed within 24 hours.

Analyze the correlation between miRNA and clinical events of cardiotoxicity, and evaluate the predictive threshold of cardiotoxicity in children with high-dose cyclophosphamide chemotherapy.Evaluate the weight of miRNA in predicting cardiac damage, combined with serum biomarkers, construct a model for Predicting the risk of myocardial damage based on speckle tracking echocardiography parameters, serum biomarkers, and miRNA expression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤14 years old;
* Bone marrow/umbilical blood HCT received high dose cyclophosphamide(>120mg/kg) ；
* ECOG≤2;
* Sign an informed consent form (<10 years old, signed by the guardian; ≥10 years old, signed by the child and guardian).

Exclusion Criteria:

* Past myocarditis, cardiomyopathy, valvular heart disease, rheumatic heart disease, severe arrhythmia, heart failure, congenital heart disease history;
* Have heart or pericardial surgery;
* Have received radiotherapy involving thoracic cavity；
* Those who do not meet the above entry criteria.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with hematopoietic stem cell transplantation received high dose cyclophosphamide(>120mg/kg)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
changes of global longitudinal strain value between cardiotoxicity group and No cardiotoxicity | From the start of cyclophosphamide injection to1 month after the completion of injection
  changes of global longitudinal strain value between cardiotoxicity group and No cardiotoxicity at the follow-up point

SECONDARY OUTCOMES:
changes of miRNA between cardiotoxicity group and No cardiotoxicity | From the start of cyclophosphamide injection to1 month after the completion of injection
  changes of miRNA between cardiotoxicity group and No cardiotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: MU Kai, Study Chair — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital (The First Affiliated Hospital of Shandong First Medical University), Jinan, Shandong, China